CLINICAL TRIAL: NCT02516631
Title: A Comparative, Open-label, Parallel Design, Bioavailability Study of Two Misoprostol Formulations (Angusta™ 25 µg Dispersible Tablets vs. Cytotec® 200 µg Tablets) Following Single Oral or Sublingual Administration and Comparison of Safety of the Two Formulations Following Repeat Dosing Until Labour
Brief Title: Comparative Bioavailability Study of Two Misoprostol Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ-201
Record Dates: First submitted 2015-06-12; First posted 2015-08-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Labour, Induced
Keywords: Labour, induced; Misoprostol; Pharmacokinetics; Cardiotocography; Safety
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral (A) (Active Comparator): One tablet of Angusta™ (25 µg) or 1/8 of a tablet of Cytotec® (25 µg).
  Interventions: Drug: Angusta™; Drug: Cytotec®
- Oral (B) (Active Comparator): Two tablets of Angusta™ 25 µg or ¼ of a tablet of Cytotec®.
  Interventions: Drug: Angusta™; Drug: Cytotec®
- Sublingual (C) (Active Comparator): Two tablets of Angusta™ (total dose of 50 µg) or ¼ of a tablet of Cytotec® (50 µg.
  Interventions: Drug: Angusta™; Drug: Cytotec®

INTERVENTIONS:
Drug: Angusta™ — One tablet of Angusta™ (25 µg) given every 2 hours
  Arms: Oral (A)
Drug: Cytotec® — 1/8 of a tablet of Cytotec® (25 µg) given every 2 hours. Drug administration should be repeated every 2 hours until labour has commenced.
  Arms: Oral (A)
Drug: Angusta™ — Two tablets of Angusta™ 25 µg given every 4 hours
  Arms: Oral (B)
Drug: Cytotec® — ¼ of a tablet of Cytotec® given every 4 hours. Drug administration should be repeated every 4 hours until labour has commenced.
  Arms: Oral (B)
Drug: Angusta™ — Two tablets of Angusta™ (total dose of 50 µg), given every 4 hours
  Arms: Sublingual (C)
Drug: Cytotec® — ¼ of a tablet of Cytotec® (50 µg), given every 4 hours. Subjects should not swallow for a period of 5 minutes. Drug administration should be repeated every 4 hours until labour has commenced.
  Arms: Sublingual (C)

SUMMARY:
The purpose of this study is to compare pharmacokinetics of two formulations of misoprostol following single dose administration in adult women being given misoprostol for cervical ripening and induction of labour.

DETAILED DESCRIPTION:
Prostaglandin E2 (dinoprostone) given vaginally or intra-cervically, and oxytocin have been the most commonly used preparations for induction of labour. Misoprostol is a synthetic prostaglandin E1 analogue. Misoprostol has anti-secretory and mucosal protective properties and was originally developed in the 1970s for the prevention of nonsteroidal anti-inflammatory drug (NSAID)-induced peptic ulcers. It is now used much more widely for 'off-label' indications like medication abortion, medical management of miscarriage, cervical ripening before surgical procedures, treatment of postpartum hemorrhage, and induction of labour. The lack of a specific license for Cytotec® to be used in obstetrics and gynecology has led to a number of problems regarding correct dose and dose regime.

The study is an open-label, randomized, single-dose, comparative, parallel design, bioavailability study followed by repeat dosing of of two formulations misoprostol in healthy adult females being induced to go into labour.

The drug shall be administered orally or sublingually.

ELIGIBILITY:
Inclusion Criteria:

* Adult females
* Women wanting to participate and having given informed consent
* Known to have reached week 37 + 0 days to week 42 + 2 days of gestation
* With a viable fetus in a vertex position
* Age above or equal to 18 years old
* Women opting for vaginal delivery
* BMI between 20 and 30 kg/m2

Exclusion Criteria:

* Women with known allergy to misoprostol or other prostaglandins
* Women with prior caesarean section
* Women with dead or anomalous fetus
* Women with twin pregnancy
* Women with known liver or renal dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) 0-t misoprostol | For 2 hours regime: pre-dose, 5, 10, 20, 30, 40, 50, 75, 100 and 120 min post-dose. For 4-hours regime at pre-dose, 5, 10, 20, 30, 40, 50, 75, 100,120, 180 and 240 min post-dose
AUC (area under the curve) 0-inf of misoprostol | For 2 hours regime: pre-dose, 5, 10, 20, 30, 40, 50, 75, 100 and 120 min post-dose. For 4-hours regime at pre-dose, 5, 10, 20, 30, 40, 50, 75, 100,120, 180 and 240 min post-dose

SECONDARY OUTCOMES:
t max (Time to maximum) of misoprostol | For 2 hours regime: pre-dose, 5, 10, 20, 30, 40, 50, 75, 100 and 120 min post-dose. For 4-hours regime at pre-dose, 5, 10, 20, 30, 40, 50, 75, 100,120, 180 and 240 min post-dose
t 1/2 (Elimination half-life) of misoprostol | For 2 hours regime: pre-dose, 5, 10, 20, 30, 40, 50, 75, 100 and 120 min post-dose. For 4-hours regime at pre-dose, 5, 10, 20, 30, 40, 50, 75, 100,120, 180 and 240 min post-dose
APGAR score of infant | At time of birth
Cardiotochographic (CTG) monitoring. | During labour
Adverse event / Serious Adverse event profile. | From screening and until 7 days post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Wide-Swensson, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital Lund, Lund, Sweden

REFERENCES:
- [Derived] Amini M, Reis M, Wide-Swensson D. A Relative Bioavailability Study of Two Misoprostol Formulations Following a Single Oral or Sublingual Administration. Front Pharmacol. 2020 Feb 12;11:50. doi: 10.3389/fphar.2020.00050. eCollection 2020. PMID 32116725